CLINICAL TRIAL: NCT06870526
Title: Program Evaluation of FOODBOX: "Feasibility of Online-supported Delivery Bringing Optimal Nutrition to Diverse Low-income Households With Children
Brief Title: Feasibility of Online-supported Delivery Bringing Optimal Nutrition to Diverse Low-income Households With Children
Acronym: FOODBOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: New York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB0010546
Record Dates: First submitted 2025-01-17; First posted 2025-03-11 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Food Insecurity
Keywords: Grocery; Food delivery

STUDY DESIGN:
Intervention Model Description: Behavioral intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FoodBox (Experimental): Participants will receive a grocery box for 12 weeks. Participants will receive groceries that contain fresh, frozen, or canned fruits, vegetables, legumes, whole grains, and low-sugar low-fat snacks.
  Interventions: Behavioral: Food box delivery

INTERVENTIONS:
Behavioral: Food box delivery — * Time Needed: 12 weeks (duration of intervention)
  * Description: Participants will receive grocery boxes containing a selection of food items tailored to their cultural and nutritional needs. They will be asked to utilize the groceries provided and provide feedback on the quality and quantity of items received. The pilot study will partner with Instacart, utilizing Instacart Care Carts for the "medically tailored grocery delivery" in which researchers order and deliver groceries on behalf of participants. Although families are not able to modify the order, they select when and where they want the grocery box delivered.

SUMMARY:
The goal of this study is to find ways to help families with children who have limited incomes get better access to healthy and culturally appropriate foods. The study will test a program called "medically tailored grocery box delivery," which sends boxes of healthy groceries to families based on their specific health needs.

The study aims to answer:

1. Can this grocery delivery program improve families' access to healthy foods and support better eating habits?
2. Will families use the groceries provided, and how effective is the program overall?

To answer these questions, researchers will:

* Work with the community to design the grocery program and make sure the foods meet families' cultural preferences.
* Test how well the program can be carried out in real-world settings.
* Compare how the program affects families' access to healthy food, eating habits, and use of the grocery boxes.

DETAILED DESCRIPTION:
The overarching goal of this project is to address nutrition insecurity among diverse low-income households with children by designing and piloting an intervention strategy grounded in Food Is Medicine (FIM). Leveraging existing online grocery technology, this project seeks to enhance nutrition security through a "medically tailored grocery box delivery" program. We aim to: 1) conduct formative research with a community engagement process to inform the intervention design and ensure foods are culturally acceptable and appropriate; 2) apply implementation strategies to assess the extent to which the intervention can be implemented in the intended setting exactly as evaluated; 3) compare preliminary efficacy of the program on nutrition security, dietary intake, and redemption rate.

Target Population: The study will be conducted in low-income, diverse neighborhoods of New York City, specifically in the South Bronx. Selection of the community was based on the highest poverty levels, chronic disease prevalence, and ethnic diversity. The target population includes households with young children (< age 10) at risk for food insecurity, primarily English or Spanish speakers, participating in SNAP or meeting income criteria < 130% FPL), and access to online ordering through a smartphone or computer.

Approach: Recruitment will be conducted at Bronx Health REACH, a community-based organization located in the South Bronx that serves residents of low-income and SNAP-eligible participants. SNAP-Ed provider and researchers will build the grocery box using Instacart. We will interview the provider to elicit barriers and opportunities for improvement and scalability of the program in other community settings. The formative research plan for the pilot study includes the incorporation of two focus groups at the beginning and end of the intervention, each comprising 10-12 participants. The pilot study will partner with Instacart, utilizing Instacart Care Carts for the "medically tailored grocery delivery" in which researchers order and deliver groceries on behalf of participants. Although families are not able to modify the order, they select when and where they want the grocery box delivered.

A total of 30 households will be selected for the program and will receive the grocery box for 12 weeks. Participants will receive groceries that contain fresh, frozen, or canned fruits, vegetables, legumes, whole grains, and low-sugar low-fat snacks. Evaluation of the intervention will encompass a comprehensive assessment of household nutrition security and dietary intake among children and caregivers. Pre- and post-assessments will evaluate household nutrition security, and diet intake among children and their caregivers using 24-hour recalls and veggie meter assessments. Additionally, SNAP-ED providers will be interviewed to gather insights into their experiences with program delivery and the utilization of Instacart for grocery box orders. A benchmark (i.e., minimum acceptable values) will be set a priori for feasibility (i.e., recruitment, randomization, intervention fidelity, and retention rates) and acceptability following the RE-AIM framework. Instacart data will track orders, deliveries, and confirmations to assess redemption rates. Acceptability will be assessed as participant satisfaction with the intervention materials. To evaluate preliminary efficacy, linear mixed-effects models with random effects to account for repeated caregiver measures will be used.

ELIGIBILITY:
Inclusion Criteria:

* Reside in low-income neighborhoods of the South Bronx, New York City.
* Have children under the age of 10 in the household.
* Primarily English or Spanish speakers.
* Participating in the Supplemental Nutrition Assistance Program (SNAP) or meeting income criteria (< 130% of the Federal Poverty Level).
* Have access to online ordering through a smartphone or computer.

Exclusion Criteria:

* Households residing outside the designated low-income neighborhoods of the South Bronx.
* No children under the age of 10 in the household.
* Unable to communicate in English or Spanish.
* Not participating in SNAP or not meeting income criteria.
* Lack access to online ordering through a smartphone or computer.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the FOODBOX pilot | 12 weeks
  Grocery Box Delivery and Usage: Participants will receive grocery boxes containing a selection of fresh, frozen, or canned fruits, vegetables, legumes, whole grains, and low- sugar, low-fat snacks. Information regarding the receipt and utilization of grocery boxes will be collected, including delivery confirmation, redemption rates, and feedback on the quality and quantity of food items received.
  Participant Feedback and Satisfaction: Participants will have opportunities to provide feedback on the intervention materials, delivery process, and overall satisfaction with the program. This feedback may be collected through surveys, interviews, or focus groups conducted at various points during the intervention period.

SECONDARY OUTCOMES:
Food Security | 12 weeks
  We will use the 18-item USDA Household Food Security Module to assess food security of families. This is a three-stage design with screeners. Screening keeps respondent burden to the minimum needed to get reliable data. Most households in a general population survey are asked only three questions (five if there are children in the household).

OTHER OUTCOMES:
Fruit and Vegetable Intake | 12 weeks
  Participants will undergo dietary intake assessments to evaluate their consumption of fruits and vegetables. In addition, participants will be assessed using a Veggiemeter by the research team, a device designed to measure vegetable intake.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Trude, PhD, Principal Investigator — New York University; Roger Figueroa Baotista, PhD, Principal Investigator — Cornell University
Locations (1):
- Bronx Health REACH, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided